CLINICAL TRIAL: NCT03459352
Title: Feasibility Study of Digital Symptom Tracking, Patient Engagement and Quality of Life in Patients Seen in GI Oncology Clinic
Brief Title: Digital Symptom Tracking, Patient Engagement and Quality of Life in GI Oncology Clinic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Noona Healthcare Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00092471
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2019-09

CONDITIONS: Cancer
Keywords: Cancer; Patient Reported Outcomes; Symptom management
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ePRO (Experimental): There is no therapeutic intervention. Patients will use ePRO system to report systems. We will describe use in patients to determine compliance in reporting symptoms.
  Interventions: Other: ePRO

INTERVENTIONS:
Other: ePRO — Patients will be instructed to log symptoms with an ePRO app using their own personal devices, and prompted once per month for 12 months to log symptoms.
  These participants will be sent an Adverse Event Questionnaire (AEQ) via the Noona tool that summarizes their symptoms and distress once per month and one week prior to any medically indicated oncology clinic visit.
  Symptoms designated as clinically severe either during regular symptom logging or via the AEQ will trigger a prompt to contact the clinical team for immediate follow-up. Participants will complete a follow-up questionnaire at 6 months and 12 months following enrollment that includes a self-report of symptom burden, HRQOL, and satisfaction.
  Other Names: Noona web-based platform

SUMMARY:
A pilot study of an ePRO system in cancer patients receiving systemic therapies.

DETAILED DESCRIPTION:
The primary purpose of this pilot study is to determine the feasibility of the Noona Healthcare Mobile PRO Application to describe oncology patient engagement using a web-based symptom self-monitoring instrument. Additionally, the studyy will dentify side effects as well as long term or chronic adverse events during and following cancer therapy based on the United States (US) National Cancer Institute (NCI) Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE), and identify patients to participate in future long-term Quality of Life studies following cancer therapy.

The study is not intended to compare outcomes between groups receiving different therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals (men and women) aged 18 years or older
2. History cancer with no limitation on prior lines of therapy in the metastatic setting
3. ECOG performance status of 0-2
4. Estimated life expectancy of at least 12 months
5. Access to smartphone, tablet or computer with capability to utilize symptom-tracking application
6. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
7. Willing and able to comply with all study procedures

Exclusion Criteria:

1. Concurrent disease or condition that interferes with participation or safety
2. Non-English speaking, as the application is developed in the English language
3. Children will not be included in the study. The pattern of disease and symptoms are different in children than in an adult population. The web-based tool was designed based on the symptom experience of adults with cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Subject participation | 12 months
  total number of subjects that participate in the use of a web-based system

CONTACTS AND LOCATIONS:
Overall Officials: H. Kim Lyerly, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States